CLINICAL TRIAL: NCT07153302
Title: Assessing Bone Fracture Healing Effect of Prunus Dulcis (Almonds) - A Randomized Controlled Trial
Brief Title: Assessing Bone Fracture Healing Effect of Almonds
Acronym: AFHEA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aga Khan University Hospital, Pakistan (Other)
Collaborators: University of Karachi (Other); PharmEvo Pvt Ltd (Industry)
Responsible Party: Principal Investigator, Zehra Abdul Muhammad, Senior Instructor, Aga Khan University Hospital, Pakistan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 58223480; 53557 (Other: The Aga Khan University)
Record Dates: First submitted 2025-08-25; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Femur Shaft Fracture; Tibia Fractures; Vitamin D; Sweet Almonds; Callus Index; Callus Bridging
Keywords: callus bridging; callus index; femur shaft fracture; tibia shaft fracture; Prunus dulcis (almonds); vitamin D3

STUDY DESIGN:
Intervention Model Description: Patients (N=136) are divided into two groups. Group 1 (vitamin D insufficiency, blood vitamin D level 21-29 ng/mL) and Group 2 (vitamin D deficiency, blood vitamin D level ≤20 ng/mL). Within two weeks of screening, patients are randomly allocated into a total of three arms.
  Note: If blood vitamin D level exceeds 50 ng/mL, the vitamin D administration will be discontinued by the trial team and treating surgeon will decide to continue it or not.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Other): Cross-over treatment
  Group 1 (N=14):
  Arm A (n=7) = 5±0.5 grams/day of whole almonds for 4 weeks, followed by 7 days washout period and initiating cross-over treatment by oral vitamin D3 200,000 units/week for 8 weeks.
  Interventions: Other: Prunus dulcis (sweet almonds)
- Arm B (Other): Cross-over treatment
  Group 1 (N=14):
  Arm B (n=7) = Oral vitamin D3 200,000 units/week for 8 weeks, followed by 7 days washout period and initiating cross-over treatment by 5±0.5 grams/day of whole almonds for 4 weeks
  Group 2 (N=122):
  Arm B (n=61) = Oral vitamin D3 200,000 units/week for 8 weeks, followed by 7 days washout period and initiating cross-over treatment by 5±0.5 grams/day of whole almonds for 4 weeks.
  Interventions: Other: Prunus dulcis (sweet almonds)
- Arm C (Other): Cross-over treatment
  Group 2 (N=122):
  Arm C (n=61) = Oral vitamin D3 200,000 units/week together with 5±0.5 grams/day whole almonds for 4 weeks, followed by 7 days washout period and initiating cross-over treatment by oral vitamin D3 200,000 units/week for 8 weeks.
  Interventions: Other: Prunus dulcis (sweet almonds)

INTERVENTIONS:
Other: Prunus dulcis (sweet almonds) — Almonds are functional food items that contain bone essential micronutrients.
  Other Names: sweet almonds

SUMMARY:
Femur and tibia shaft fractures are common after trauma with a burden of 5% and 20% respectively. Clinicians recommend costly bone strengthening drugs/supplements while treating bone fractures. These drugs have side effects and are costly due to which patients skip these supplements. Routinely prescribed vitamin D have known toxicity. To overcome this problem, affordable and safe alternative treatment is needed. Sweet almonds contain essential bone nutrients that might have potential for maintaining bone strength. Human and animal studies have shown positive impact of almonds on bone health and fracture healing. Almonds are consumed in diet frequently but may occasionally cause toxicity, mainly if consumed at higher amount. Because of the high bone essential nutrients in almonds, the trial aimed to investigate the fracture healing effect and safety of almonds in femur and tibia shaft fractures. This might provide an alternate option for bone supplants while treating fractures.

Hypothesis: Compared to routine vitamin D3, almonds non-inferiorly improves fracture callus index and raise vitamin D3 level in blood in femur and tibia shaft fracture patients.

Primary Objectives:

1. To compare tibia and femur shaft fracture callus index and callus bridging on x-rays at 4 and 13 weeks herewith group 1 suffering vitamin D insufficiency (arm A versus arm B) and group 2 suffering vitamin D deficiency (arm B versus arm C) treated as cross-over with oral whole almonds and vitamin D3.
2. To compare the incidence of adverse events between almonds and vitamin D3 treatments up to 13 weeks follow-up.

Secondary Objectives:

1. To compare the almonds and vitamin D3 treatment cost.
2. To compare within group blood vitamin D levels (ng/mL) at baseline and post-treatment follow-ups.

Methods:

Study design: Single-center, open-labeled, crossover, non-inferiority randomized controlled trial.

Total 136 subjects are required with 14 subjects in group 1 and 122 in group 2.in 24-month duration.

Study procedures:

1. Regulatory and Ethical approvals.
2. Patient screening and eligibility assessment. Patients, of 18 to 55 years of age of any gender, with trauma associated femur and tibia shaft fractures who agree to voluntary participate are included and mentally retarded or patients with severe psychiatric illness, already on or require bone-strengthening drugs , having severe cardiovascular, hepatic, or renal disease, known allergy/toxicity to almonds and/or vitamin D supplements.
3. Written informed consent administration.
4. Randomization Patients (N=136) are divided into two groups. Group 1 (N=14, vitamin D insufficiency, blood vitamin D level 21-29 ng/mL) and Group 2 (N=122, vitamin D deficiency, blood vitamin D level ≤20 ng/mL).

   I. Group 1 (N=14):

   Arm A (n=7)=5 grams/day of almonds for 4 weeks, followed by 7 days washout period and cross-over treatment by oral vitamin D3 200,000 units/week for 8 weeks.

   Arm B (n=7)=Oral vitamin D3 200,000 units/week for 8 weeks, followed by 7 days washout period and cross-over treatment by 5 grams/day of almonds for 4 weeks

   II. Group 2 (N=122):

   Arm B (n=61)=Oral vitamin D3 200,000 units/week for 8 weeks, followed by 7 days washout period and cross-over treatment by 5 grams/day of almonds for 4 weeks.

   Arm C (n=61)=Oral vitamin D3 200,000 units/week together with 5 grams/day almonds for 4 weeks, followed by 7 days washout period and cross-over treatment by oral vitamin D3 200,000 units/week for 8 weeks.
5. Patients are followed at 4 weeks and 13 weeks follow-ups after treatment.
6. Fracture site routine X-rays and RUST scores are assessed by treating surgeon/investigator(s) at follow-ups for bone fracture healing.
7. Investigational product (IP) safety assessment and reporting as per ICH-GCP guidelines. Subjects experiencing any adverse event (AE)/serious adverse event (SAE) is provided optimum care at earliest. All relevant reporting bodies are notified within recommended timeline.
8. The almonds are regularly purchased from the Purchase Department of the Hospital, weighted, packaged and labelled, and stored at the secure dry hygienic place. The product is dispensed to the patient and a daily IP diary is provided for compliance.
9. Patients can withdraw from the study at any time without losing any of his/her patient rights.
10. Study close-out process will be of one to two-month duration.

Statistical analysis:

The SPSS version 19.0 will be used to analyze data. Quantitative variables will be expressed as mean±SD/median (IQR) and qualitative as frequencies (%). IP related AEs/SAEs will be assessed by incidence/stratification. Witin group and within arm comparisons for the radiological assessments and vitamin D3 level will be analyzed by ANOVA and GEE. Within arm tibia and femur fracture outcomes will be compared by independent t-test/Mann Whitney U test. The p-value <0.05 is considered significant. Multiple regression analysis for association of covariates and outcome will be used.

DETAILED DESCRIPTION:
Trauma is a leading cause of morbidity and mortality in low middle income countries with road traffic accident as a common mechanism of trauma. Femur and tibia shaft fractures are common with a burden of 5% and 20% respectively. For proper fracture healing and treatment, vitamin D supplements are prescribed in routine practice. Vitamin D can cause confusion, polyuria, thirst, anorexia, vomiting, constipation, nausea, arrhythmias, seizures, potentiate cardiac drugs, renal failure, tissue calcium deposit, bone demineralization, muscle/bone pain, allergy, weakness, metallic taste, weight loss, chest pain, dyspnea. In developing countries, most patients skip supplements due to the unaffordability, toxicity, and inaccessibility of slums. Considering the vitamin D cost and toxicity, alternative effective, safe, and affordable treatment is a prerequisite. Prunus dulcis (sweet almonds) is a dietary item which contains essential bone micronutrients that contribute in bone health for structural strength and proper functioning. evidence shows enormous health benefits of almonds According to one study, 60 grams of Prunus dulcis (almonds) reduced osteoclast formation and calcium release, indicating a positive effect on bone health. In another study, Prunus dulcis extract accelerated tibial bone fracture healing in rabbits, which is another evidence for potential benefits of Prunus dulcis on bone healing and health. In continuation to this, other health benefits are also reported. Prunus dulcis (almond) are consumed as a dietary item but it may occasionally cause allergy and if consumed in higher amount (~11 grams/day), can cause toxicity Based on the available facts, the current trial question is whether addition of Prunus dulcis (almonds) in the diet is safe, assists fracture healing, and improve vitamin D levels in blood in the femur and tibia shaft fractures compared to routine vitamin D supplement? It is hypothesized that compared to routine vitamin D3, Prunus dulcis (almonds) non-inferiorly improves fracture callus index with raise in vitamin D3 level in blood in femur and tibia shaft fracture patients.

The clinical trial aims to evaluate and compare the safety and effect of Prunus dulcis (almonds) on callus formation and callus bridging in femur and tibia shaft fractures and improvement in vitamin D level in blood up to 13 weeks compared to routine vitamin D supplements. This might assist orthopaedic surgeons in optimizing bone healing through almonds in patients arriving with fracture injuries as an alternative dietary bone nutritive source.

Primary Objectives:

3. To compare tibia and femur shaft fracture callus index (mm) and callus bridging (The Radiological Union Score for Tibial fractures-RUST) on x-rays at 4 and 13 weeks herewith group 1 suffering vitamin D insufficiency (arm A versus arm B) and group 2 suffering vitamin D deficiency (arm B versus arm C) treated as cross-over with oral 5 grams/day whole almonds and 200,000IU/week vitamin D3.

4. To compare the incidence of adverse events between almonds and vitamin D3 treatments in all trial arms up to 13 weeks follow-up.

Secondary Objectives:

3. To compare the average almonds and vitamin D3 treatment cost. 4. To compare within group blood vitamin D levels (ng/mL) at baseline and post-treatment at 4 and 13 weeks.

Methods:

Number of participants: 136 Study design: Single-center, open-labeled, crossover (1:1 for each group), non-inferiority randomized controlled trial.

Study Duration: 24 months

Study procedures:

After Institutional and Ethical Review Committee approvals, patient eligibility is assessed by the designated trained researcher in in-patient and outpatient orthopaedic units.

Consent administration process: Informed written consent (English and Urdu) administration as per Good Clinical Practice Guidelines (GCP) guidelines. Clinical trial method is explained to patients. Patients are allowed to read the consent form and ask questions. A signed consent copy is provided to each subject.

Patient Screening:

Eligibility criteria: assessment. Sampling Method: Non-probability, consecutive sampling

Randomization:

Patients (N=136) are divided into two groups. Group 1 (vitamin D insufficiency, blood vitamin D level 21-29 ng/mL) and Group 2 (vitamin D deficiency, blood vitamin D level ≤20 ng/mL). Within two weeks of screening, patients are randomly allocated into a total of three arms.

III. Group 1 (N=14):

Arm A (n=7) = 5±0.5 grams/day of whole almonds for 4 weeks, followed by 7 days washout period and initiating cross-over treatment by oral vitamin D3 200,000 units/week for 8 weeks.

Arm B (n=7) = Oral vitamin D3 200,000 units/week for 8 weeks, followed by 7 days washout period and initiating cross-over treatment by 5±0.5 grams/day of whole almonds for 4 weeks

IV. Group 2 (N=122):

Arm B (n=61) = Oral vitamin D3 200,000 units/week for 8 weeks, followed by 7 days washout period and initiating cross-over treatment by 5±0.5 grams/day of whole almonds for 4 weeks.

Arm C (n=61) = Oral vitamin D3 200,000 units/week together with 5±0.5 grams/day whole almonds for 4 weeks, followed by 7 days washout period and initiating cross-over treatment by oral vitamin D3 200,000 units/week for 8 weeks.

Patient follow-ups and Data Collection:

Patients are followed at 4 weeks±1 week and 13 weeks±1 week follow-up visits after treatment. In order to reduce bias, researchers were trained on data collection form and GCP guidelines prior to data collection. In case of lost to follow-up, patients are contacted by telephone to gather necessary information.

Assessments:

Fracture site routine X-rays and RUST score for bone fracture healing are assessed by treating surgeon/investigator(s) at follow-ups.

The research study does not seem to have any potential health hazard as vitamin D is routinely prescribed, and almonds are consumed as a dietary item. Complying with all regulatory standards and as per International Conference on Harmonisation of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH) Good Clinical Practice (GCP) guidelines, study subjects experiencing any adverse event (AE)/serious adverse event (SAE) will be provided optimum care at earliest. Principal Investigator is responsible for sending reports to the reporting bodies (Ethical Review Committee, Sponsor etc.) as required.

Investigational product handling: The investigational products is regularly purchased from the Purchase Department of the Hospital, weighted, packaged, and properly labelled by the designated researcher and stored at the secure dry hygienic place. The product is dispensed to the patient by the designated researcher. The daily diary is provided to the patients for compliance and investigational product intake. The returns of used packs/products are collected at follow-ups.

Data management:

Data is managed at the Department of Surgery. Randomization list is generated. Data is kept secure in cabinets with a lock and key and a password-protected system with controlled data access. Fifteen percent of the data is double-checked/validated by the Principal Investigator. Data will be archived and stored for 15 years or longer after study completion.

Statistical Consideration:

The Statistical Package for Social Sciences (SPSS) version 19.0 will be used to analyze data. Quantitative variables (age, callus index, vitamin D3 level, etc.) will be expressed as mean±SD or median (IQR) as appropriate and qualitative variables (gender, type of fracture, etc.) as frequencies (percentages). Data will be analyzed by intention to treat analysis. Investigational product related AEs/SAEs will be assessed by incidence and stratification. Per group between arms comparisons for the mean difference of callus index, RUST scores, and vitamin D3 level will be analyzed by mixed ANOVA and within arms follow-up observation by repeated measures ANOVA/Freidman test and generalized estimating equation (GEE). Femur and tibia fractures within each arm will be compared for callus index and vitamin D levels by independent student t-test/Mann Whitney U test (as appropriate). The p-value less than 0.05 will be considered statistically significant with a confidence interval of 95%. Multiple regression will be used to assess the association between covariates like age, gender, fracture type, etc., and a numeric outcome like callus index, vitamin D3 level, etc. The percentage of lost to follow-ups will also be assessed.

Withdrawals: Patients can withdraw from the study at any time without losing any of his/her patient rights.

Study Close-out:

Study close-out process will be of one to two-month duration.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of 18 to 55 years of age of any gender.
2. Agree and able to voluntary participate.
3. Patients with trauma associated femur fracture and tibia shaft fracture arriving at hospital for treatment.

Exclusion Criteria:

1. Mentally retarded or patients with severe psychiatric illness.
2. Patients are already on bone-strengthening drugs (bisphosphonates, vitamin D, strontium ranelate, teriparatide, etc.).
3. Patients who require bone-strengthening drugs for osteoporosis or for any urgent need.
4. Severe cardiovascular, hepatic, or renal disease.
5. Known allergy or toxicity to Prunus dulcis (almonds) and/or vitamin D supplements.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Callus index | comparable callus formation at 4 and 13 weeks post-treatment.
  Assessing mean difference in femur and tibia shaft fracture bone callus formation by measuring callus index (millimetre diameter) on x-ray (AP and ML/Lateral views) at follow-ups post-treatment. Callus index is defined as the ratio of the maximum callus diameter to bone diameter at the same level as the callus. Callus index determined for anteroposterior (AP) and mediolateral (ML) radiographs.
Callus bridging | Comparable callus bridging at 4 and 13 weeks post-treatment,
  Callus bridging on x-ray (AP and ML/Lateral views) at follow-ups post-treatment, the fracture heals by a periosteal bony callus at the periphery of the fracture and fibrocartilaginous bridging callus between bone ends. Radiographic union scale in tibial fractures (RUST) score standardize the radiographic assessment of tibial fractures by assessing cortical bridging and obliteration of fracture line. A RUST score of 1 (cortex with no callus and a visible fracture line), 2 (a bridging callus and a visible fracture line); and 3 (a callus and no visible fracture line). Low RUST score (4 or 5) indicates no or poor fracture healing. High score (11 or 12) indicates definite fracture healing.
Investigational product safety | Fifty percent fewer side effects after almonds than vitamin D3 treatments. SAE within 24 hours unexpected AE 15 days of knowing the event, SAE report submission within 5 days and unexpected AE in 15 days.
  Assessment of patient safety of all three treatment arms by serious adverse event (SAE)/adverse event (AE) incidence. Any untoward medical occurrence in a patient administered a medicinal product is called an AE. If any dose results in death, disability/incapacity, inpatient/prolonged hospitalization, and is life-threatening is called an SAE.

SECONDARY OUTCOMES:
Blood Vitamin D level | Blood vitamin D3 levels comparable after 28 days of almonds and 8 weeks after routine vitamin D3 treatments with one week washout time.
  Assessing mean raise in vitamin D ng/mL level in blood after almonds and routine vitamin D3 treatments. Vitamin D3 insufficiency is 21-29 ng/mL while deficiency is 20 ng/ml or below.
Cost | Almonds cost 28 days of treatment and vitamin D cost 8 weeks of treatment.
  Low average cost of almonds treatment compared to vitamin D supplements.

CONTACTS AND LOCATIONS:
Overall Officials: Zehra A Muhammad, M.B.B.S., M.S. Research, Principal Investigator — Aga Khan University
Locations (1):
- The Aga Khan University, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data on demographics, outcome, SAE/AE.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After study close-out and on request.
Access Criteria: At the time of publication (deidentified individual patient data and analysis plan) and on request after study close-out (Study protocol, clinical study report).

REFERENCES:
- [Background] Barreca D, Nabavi SM, Sureda A, Rasekhian M, Raciti R, Silva AS, Annunziata G, Arnone A, Tenore GC, Suntar I, Mandalari G. Almonds (Prunus Dulcis Mill. D. A. Webb): A Source of Nutrients and Health-Promoting Compounds. Nutrients. 2020 Mar 1;12(3):672. doi: 10.3390/nu12030672. PMID 32121549
- [Background] Leow JM, Clement ND, Tawonsawatruk T, Simpson CJ, Simpson AH. The radiographic union scale in tibial (RUST) fractures: Reliability of the outcome measure at an independent centre. Bone Joint Res. 2016 Apr;5(4):116-21. doi: 10.1302/2046-3758.54.2000628. PMID 27073210
- [Background] Whelan DB, Bhandari M, Stephen D, Kreder H, McKee MD, Zdero R, Schemitsch EH. Development of the radiographic union score for tibial fractures for the assessment of tibial fracture healing after intramedullary fixation. J Trauma. 2010 Mar;68(3):629-32. doi: 10.1097/TA.0b013e3181a7c16d. PMID 19996801
- [Background] Eastaugh-Waring SJ, Joslin CC, Hardy JR, Cunningham JL. Quantification of fracture healing from radiographs using the maximum callus index. Clin Orthop Relat Res. 2009 Aug;467(8):1986-91. doi: 10.1007/s11999-009-0775-0. Epub 2009 Mar 13. PMID 19283438
- [Background] Anaraki N, Beyraghi AH, Raisi A, Davoodi F, Farjanikish G, Sadegh AB. The effect of aqueous extract of Prunus dulcis on tibial bone healing in the rabbit. J Orthop Surg Res. 2021 Jun 7;16(1):362. doi: 10.1186/s13018-021-02498-z. PMID 34098995
- [Background] Platt ID, Josse AR, Kendall CW, Jenkins DJ, El-Sohemy A. Postprandial effects of almond consumption on human osteoclast precursors--an ex vivo study. Metabolism. 2011 Jul;60(7):923-9. doi: 10.1016/j.metabol.2010.08.012. Epub 2010 Oct 13. PMID 20947104
- [Background] Jamshed H, Arslan J, Sultan FT, Siddiqi HS, Qasim M, Hassan Gilani AU. Almond protects the liver in coronary artery disease: A randomized controlled clinical trial. J Pak Med Assoc. 2021 Mar;71(3):791-795. doi: 10.47391/JPMA.198. PMID 34057922
- [Background] Jalali-Khanabadi BA, Mozaffari-Khosravi H, Parsaeyan N. Effects of almond dietary supplementation on coronary heart disease lipid risk factors and serum lipid oxidation parameters in men with mild hyperlipidemia. J Altern Complement Med. 2010 Dec;16(12):1279-83. doi: 10.1089/acm.2009.0693. Epub 2010 Nov 29. PMID 21114415
- [Background] Zofkova I, Nemcikova P, Matucha P. Trace elements and bone health. Clin Chem Lab Med. 2013 Aug;51(8):1555-61. doi: 10.1515/cclm-2012-0868. PMID 23509220
- [Background] Myung SK, Kim HB, Lee YJ, Choi YJ, Oh SW. Calcium Supplements and Risk of Cardiovascular Disease: A Meta-Analysis of Clinical Trials. Nutrients. 2021 Jan 26;13(2):368. doi: 10.3390/nu13020368. PMID 33530332
- [Background] Fischer V, Haffner-Luntzer M, Amling M, Ignatius A. Calcium and vitamin D in bone fracture healing and post-traumatic bone turnover. Eur Cell Mater. 2018 Jun 22;35:365-385. doi: 10.22203/eCM.v035a25. PMID 29931664
- [Background] Doetsch AM, Faber J, Lynnerup N, Watjen I, Bliddal H, Danneskiold-Samsoe B. The effect of calcium and vitamin D3 supplementation on the healing of the proximal humerus fracture: a randomized placebo-controlled study. Calcif Tissue Int. 2004 Sep;75(3):183-8. doi: 10.1007/s00223-004-0167-0. PMID 15386160
- [Background] Brun-Buisson C. [Treatment of antibiotic-resistant bacteria at the intensive care unit: a therapy dilemma]. Int J Clin Pract Suppl. 2000 Jan;(109):4-5. No abstract available. Italian. PMID 10765553